CLINICAL TRIAL: NCT05821270
Title: Effects of Ashtanga-Vinyasa Yoga Supta on Portuguese Airforce Military Pilots Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Sara Alexandra Goncalves Santos, Principal Investigator, University of Évora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UEvora approval number: 21050
Record Dates: First submitted 2023-02-08; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Military Operational Stress Reaction
Keywords: yoga; airforce pilots; operational performance; military pilots

STUDY DESIGN:
Intervention Model Description: 1 group randomly divided in: yoga intervention plus regular military training; and "waiting list" with only military training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): Yoga practice: 12-week program of Ashtanga Vinyasa Yoga Supta for 1h twice a week
  Interventions: Other: Ashtanga Vinyasa Yoga Supta
- Waiting list (No Intervention): Only mandatory pilot trainig that everyone in the academy receives

INTERVENTIONS:
Other: Ashtanga Vinyasa Yoga Supta — Ashtanga (asta - eight, anga - parts); Vinyasa (freely sequenced practice); Yoga (practice for evolution); Supta (closed eyes)
  Other Names: Yoga class
  Arms: Yoga

SUMMARY:
A total of 18 military pilots in their tirocinium in the air force academy from the Portuguese Air Force course "Masters in Military Aeronautics: aviator pilot specialist" participated in this study. Participants were randomly assigned to yoga (intervention group) or waiting list (control group). Procedures were approved by the Évora University research ethics committee and participants will give written informed consent according to the Helsinki declaration (approval number: 21050).

DETAILED DESCRIPTION:
A randomized, prospective, controlled trial was designed, with the participants (n=18) randomly distributed into two groups. The Control Group (n=8) will be receiving the protocolized classes from the course "Masters in Military Aeronautics: aviator pilot specialist" for 12 weeks, the Intervention Group (n=10) will receive the same course and 2 sessions per week (1h each) of the yoga classes (4). The intensity of the program (Borg rating of perceived exertion scale) will be measured. The operative performance response measurements will be collected at baseline and post-intervention. Participants will complete the following emergency protocols in a flight simulator: (1) take-off engine failure, (2) flight engine failure close to the base, (3) flight engine failure far away from the base, and (4) alternator failure. This intervention protocol was accepted by the Portuguese Airforce to be applied on Airbase 11 in Beja.

ELIGIBILITY:
Inclusion Criteria:

* healthy military pilots in their tirocinium in the air force academy from the Portuguese Air Force course "Masters in Military Aeronautics: aviator pilot specialist

Exclusion Criteria:

* military pilots on active duty before or after the tirocinium;
* injured military pilots;
* military pilots on sudden lifestyle changes (as in: starting or quitting smoking habits; starting or quitting any kind of medication; starting a new diet)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Operative performance | measured at 12 weeks (versus baseline values)
  Flight times to complete tasks in the flight simulator and report from the flight simulator controler
Changes in Stress and HRV | measured at 12 weeks (versus baseline values)
  Heart rate variability measured with Polar H10 portable device
Changes in Vestibular system control responses | measured at 12 weeks (versus baseline values)
  Postural control responses through CoP displacement measured with a portable force platform Biosignals Plux with data sampled at 1000 Hz and electrode impedance below 5 kΩ. Preprocessing performed using the EEGLAB toolbox, which is available for use in MATLAB (The MathWorks Inc., Natick, MA). Data downsampled to 100 Hz.

SECONDARY OUTCOMES:
Changes in Body composition | measured at 12 weeks (versus baseline values)
  Body composition data (percent body fat, percent fat free mass, percent muscle mass index, as a percentages) measured with a Tanita (MC-780 MA, Tanita, Tokyo, Japan) to get a bioelectrical impedance analysis (BIA) will indicate if the exercise protocol had any impact in the pilot's physical makeup.
  Percent body fat, percent fat-free mass, and percent muscle mass index are all related to body composition. Here's how they relate to each other: Percent body fat is the percentage of body weight that is made up of fat and includes both essential and storage fat; Percent fat-free mass is the percentage of body weight that is not fat and includes muscle, bone, organs, and other non-fat tissues; Percent muscle mass index is the percentage of body weight that is muscle. Percent body fat and percent fat-free mass are complementary measures that add up to 100%, while percent muscle mass index is a measure of the proportion of muscle in the body weight.
Changes in Lung capacity | measured at 12 weeks (versus baseline values)
  Ventilatory response measured with spirometry - FEV1/FVC ratio indicates how much air you can forcefully exhale
Five Facet Mindfulness Questionnaire - Changes in cognitive habilities | measured at 12 weeks (versus baseline values)
  FFMQ with 15 questions and average scores are calculated by summing the responses and dividing by the number of items, and indicate the average level of agreement with the each subscale (1 = rarely true, 5 = always true). Higher scores are indicative of someone who is more mindful in their everyday life.
Multidimensional Assessment of Interoceptive Awareness Questionnaire - Changes in cognitive habilities | measured at 12 weeks (versus baseline values)
  MAIA - is an 8-scale state-trait questionnaire with 32 items to measure multiple dimensions of interoception; scores are between 0 and 5, where higher score equates to more awareness of bodily sensation.
Aviation Safety Attitude Scale - Changes in cognitive habilities | measured at 12 weeks (versus baseline values)
  ASAS - consists of. 27 items on a five-point scale, each designed specifically to assess pilots' attitudes with respect to predict the hazardous event involvement of aviators; For all the attitude subscales, higher scores indicate a greater degree of that particular attitude - For example, higher scores on the ASAS self-confidence factor indicated that the person expressed greater confidence in their ability as a pilot

CONTACTS AND LOCATIONS:
Overall Officials: Sara G Santos, Principal Investigator — University of Évora
Locations (1):
- UEvora, Evora, Portugal

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2023 onwards
Access Criteria: Depends on the Journal that publishes the data

REFERENCES:
- [Derived] Santos S, Villafaina S, Parraca JA, Fernandes O, Melo F. The Impact of Yoga Practice on Health, Strength, and Respiratory Capacity in Portuguese Airforce Pilots: an Applied Psychophysiology and Biofeedback Approach. Appl Psychophysiol Biofeedback. 2025 Jun 13. doi: 10.1007/s10484-025-09719-9. Online ahead of print. PMID 40512335
- [Derived] Santos S, Melo F, Fernandes O, Parraca JA. The effect of Ashtanga-Vinyasa Yoga method on air force pilots' operational performance. Front Public Health. 2024 May 1;12:1334880. doi: 10.3389/fpubh.2024.1334880. eCollection 2024. PMID 38751579